CLINICAL TRIAL: NCT00249314
Title: A Prospective, Cross-Sectional, Case-Control, Molecular Study of Health Assessment and Risk in Ethnic Groups
Brief Title: (Mol-SHARE) Molecular Study of Health Assessment and Risk in Ethnic Groups
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Organization: McMaster University (Other)
Other Study IDs: Mol-SHARE
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Insulin Resistance; Type 2 Diabetes Mellitus; Cardiovascular Diseases
Keywords: South Asians; European Caucasians; ethnic differences; body composition; body fat distribution; adipose tissue; visceral fat; myocellular lipids; skeletal muscle
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to directly compare the body composition, body fat distribution, and morphological and functional features of adipose tissue and skeletal muscle between South Asians and European Caucasians.

DETAILED DESCRIPTION:
Excess body fat, the hallmark of obesity is a major risk factor for the development of insulin resistance (decreased insulin sensitivity), type 2 diabetes, and cardiovascular disease. Previous studies have shown that South Asians (people who originate from the Indian subcontinent) appear particularly prone to develop diabetes and heart disease compared to white Caucasians of European origin. In Canada, in the Study of Health Assessment and Risk in Ethnic groups (SHARE), it was observed that in a random selection of South Asian and European individuals, South Asians had twice as much type 2 diabetes and cardiovascular disease and were significantly more insulin resistant than Europeans despite a similar body mass index (BMI) and waist circumference. It is possible that the increased propensity of South Asians to develop insulin resistance, type 2 diabetes, and cardiovascular disease is related to greater total body fat and/or increased visceral fat in addition to the possible biological differences in adipose tissue and skeletal muscle tissues. The primary objective of this study is therefore to determine differences among age, sex, and BMI-matched people of South Asian and European Caucasian descent in body composition (specifically total body fat, lean body mass) and fat distribution (where the fat is stored in the body). This study will therefore test the hypothesis that for a similar BMI, South Asians have more total body fat and less lean body mass than age and sex-matched European Caucasians. The secondary objectives of this study are to look at the differences in the two ethnic groups at a biological level, including: differences in visceral fat, adipose tissue morphology, imflammation and adipokine production, skeletal muscle fat content, fatty acid oxidation and mitochondrial activity.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Between 18-50 years of age
* Fits into one of the following BMI-Strata:

  * Stratum 1: BMI 18.5 - 25 kg/m2
  * Stratum 2: BMI 25.1 -29.9 kg/m2
  * Stratum 3: BMI 30 -45 kg/m2
* Ability and willingness to complete dietary and activity diaries and questionnaires

Exclusion Criteria:

* Concurrent antidiabetic, antithypertensive, antiobesity or lipid-lowering medication
* Use of systemic glucocorticosteroids (topical and inhaled corticosteroids are acceptable)
* If the participant has any one or more of the following medical disorders:

  * Known Diabetes
  * Known renal impairment
  * Known uncontrolled endocrine disorder (e.g. hyperthyroidism, Cushing's syndrome, acromegaly, etc.)
  * Recent (less than three months) major surgery or hopitalization for severe illness
  * History of active malignancy, chronic inflammatory disorder, or chronic infections which would interfere with the protocol completion
  * Any other medical, social or geographic condition, which in the opinion of the investigator would not allow safe or reliable completion of the protocol
* Anticoagulant therapy (e.g. Coumadin)
* Orthopaedic contraindication to exercise test
* Significant fluctuations in weight over past 3 months (e.g. >10%)
* Extreme weight loss diets (e.g. Atkins, Bernstein)
* History of drug or alcohol dependency within six months prior to signing the informed consent form
* If the participant has any contraindications to MRI:

  * If the participant is clautrophobic or suffers from fear of closed spaces
  * If participant has had significant contact with metal (e.g. welding)
  * If participant has foreign body in their eye as confirmed by X-ray of the orbits
  * Body Mass Index > 45 kg/m2
  * Participant has had hip or joint replacement surgery 6-8 weeks prior to start of study
  * If participant has:

    * Cardiac pacemaker
    * Artificial cardiac valve
    * Aneurysm clip
    * Neurostimulator
    * Other implanted devices or metal objects in their body

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120
Dates: Start 2005-11; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Arya M Sharma, MD, FRCPC, Principal Investigator — McMaster University; Sonia Anand, MD, FRCPC, Principal Investigator — McMaster University; Mark Tarnopolsky, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences - Cardiovascular Obesity Research and Management Center, Hamilton, Ontario, Canada